CLINICAL TRIAL: NCT06206915
Title: To Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of XZ120 in Patients With Malignant Tumors in a Phase Ⅰ Clinical Trial
Brief Title: Phase I Study of XZ120 in Malignant Tumors
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shandong New Time Pharmaceutical Co., LTD (Industry)
Collaborators: Fudan University (Other); Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NTP-XZ120-001
Record Dates: First submitted 2023-12-20; First posted 2024-01-16 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2023-12

CONDITIONS: Advanced Malignancies

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- XZ120 monotherapy (Experimental)
  Interventions: Drug: XZ120 injection

INTERVENTIONS:
Drug: XZ120 injection — in Part One：XZ120 monotherapy, IV, no less than 60min, Q3W dose escalation study: 4 dose group (0.75 mg/m2, 1.5 mg/m2, 2.25 mg/m2, 3.0 mg/m2) Dose expansion study: MTD dose

SUMMARY:
This research includes two parts: the first part of the patients with late malignant tumor monotherapy study, at the beginning of the second part in treat DLBCL and research on combination therapy in patients with advanced breast cancer.

Research purpose: to evaluate XZ120 safety, tolerability, for the treatment of malignant tumor patients pharmacokinetic characteristics and preliminary effectiveness.

ELIGIBILITY:
Inclusion Criteria:

1. male or female aged ≥18 years old;
2. The enrolled population was divided into the first part of monotherapy and the second part of combination therapy:

   The first part of the monotherapy study was as follows:

   A: single drug dose escalation is confirmed by histology and cytology and received a standard after treatment failure or intolerance to standard treatment or for other reasons can not accept standard or the lack of effective treatment of patients with late malignant tumor; B:Single-agent dose expansion: patients with histologically or cytologically confirmed advanced breast cancer who are eligible for standard anthracycline monotherapy;

   The second part of the combination therapy dose expansion phase consists of the following cohorts:

   Cohort 1: the pathology diagnosed patients with DLBCL treated first; Cohort 2: Histologically or cytologically confirmed advanced breast cancer patients eligible for anthracycline-based standard therapy;

   Note: The patients with advanced breast cancer met any of the following criteria: ① Initially diagnosed as inoperable locally advanced or metastatic breast cancer; (2) did not receive chemotherapy after the eradicative resection of recurrent or metastatic breast cancer; ③ Recurrent or metastatic breast cancer after receiving anthracyclines for more than 12 months;
3. subjects with at least one measurable and evaluable target lesion were enrolled in the dose-expansion phase;
4. patients with ECOG performance status score of 0-1;
5. dose extension stage lymphoma patients international prognostic index (IPI) score of 0 ~ 2 points;
6. the researchers determine subjects were expected to survive a period of 3 months or more;
7. heart echocardiography measured LVEF 50% or higher;
8. important organ function meet the following requirement (first dose not allowed within 2 weeks before blood transfusion treatment, and use the growth factors of drug) : Blood routine: absolute neutrophil count (ANC) ≥1.5×109/L; The platelet count 75 x 109 / L or higher; Hemoglobin (Hb) ≥90g/L; Liver function: aspartate aminotransferase (AST), alanine aminotransferase (ALT) ≤2.5×ULN, total bilirubin (TBIL) ≤1.5×ULN; If there is liver metastasis, AST and ALT≤5×ULN, TBIL≤3×ULN; Renal function: serum creatinine (Cr) <1.5×ULN or creatinine clearance ≥50mL/min (Cr≥1.5×ULN); coagulation function: international standardization ratio (INR) 1.5 x ULN or less and part activated clotting time (APTT) live enzymes acuities were 1.5 x ULN;
9. understand the procedure and content of the trial and sign the informed consent form voluntarily.

Exclusion Criteria:

1. always use too much Doxorubicin (or pirarubicin) > total cumulative dose of 360 mg/m2, or epirubicin total cumulative quantity > 600 mg/m2;
2. patients received antineoplastic therapy 4 weeks before the first dose or within 5 half-lives of the drug, whichever was less; Patients who received a modern traditional Chinese medicine preparation with anti-tumor effect approved by NMPA within 2 weeks before the first medication;
3. Prednisone acetate tablets at a maximum dose of >100mg or equivalent cortisol for more than 5 days for the purpose of controlling lymphoma symptoms in patients with lymphoma; For other purposes, use of prednisone acetate tablets at a dose of >30mg per day or a cortisol equivalent for more than 10 days (for patients receiving ≤30mg per day of prednisone acetate tablets or a cortisol equivalent, there was a written record of stable use of the dose for at least 4 weeks before randomization);
4. patients with high-grade B-cell lymphoma;
5. the toxicity of previous antineoplastic therapy has not recovered to ≤ grade 1 according to CTCAE version 5.0 definition (except alopecia);
6. patients with other malignant tumors within 5 years before enrollment, except for the following: (1) radical cervical carcinoma in situ or non-melanoma skin cancer; (2) second primary cancer after radical resection without recurrence within 5 years; (3) The investigators thought that both patients with double primary cancers might benefit from this study; (4) if the metastatic lesion was clearly excluded from the primary tumor;
7. primary central nervous system (CNS) malignant tumor, CNS metastasis failed by local treatment, and carcinomatous meningitis; Patients with asymptomatic brain metastases or clinically stable neurological symptoms and no need for steroids and other treatments for brain metastases for more than 4 weeks were eligible for enrollment.
8. patients with a history of organ or allogeneic bone marrow transplantation or autologous stem cell transplantation within 3 months before the first dose;
9. patients who underwent major surgery within 4 weeks before the first dose or minor surgery within 2 weeks before the first dose or who have not recovered from surgery (excluding diagnostic surgery);
10. hepatitis b: HBsAg positive and/or HBcAb positive, and HBV DNA drop degree is higher than 2000 iu/mL or 104 copies/mL (hepatitis b virus infection should receive antiviral treatment according to local standard treatment guidelines and willing to accept the antiviral treatment) during the whole research; C: HCV antibody positive, and HCV RNA upper limit of normal value is higher than research center;
11. human immunodeficiency virus antibody (Anti-HIV) positive and active syphilis infection;
12. patients with uncontrolled or severe cardiovascular disease, congestive heart failure (NYHA class Ⅱ or above), unstable angina pectoris, myocardial infarction and other cardiovascular diseases within 6 months before the first drug administration; Patients with uncontrolled hypertension (systolic blood pressure ≥180mmHg and/or diastolic blood pressure ≥100mmHg);
13. has the following patients medical history, including but not limited to active autoimmune diseases, active infection (such as active tuberculosis), severe mental illness, serious endocrine diseases such as serious abnormal thyroid function;
14. for the first time to give medicine have received within 4 weeks before any other clinical trial drug/instruments treatment;
15. with a history of drug abuse or alcohol abuse within 6 months before the first drug administration;
16. patients with a history of severe allergy or known previous allergy to anthracyclines or anthradiones, or to any component of the investigational drug;
17. planning to receive live or live attenuated vaccine within 4 weeks before the first dose or during the study;
18. pregnancy or lactation women, women of childbearing age subjects or partner for women of child-bearing age male subjects to study period, and at the end of the study medication use medical certification within six months after effective contraceptive measures (such as intrauterine device or a condom);
19. the researchers determine doesn't fit into the group.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2025-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
The incidence of XZ120 treatment-emergent adverse events | 36 courses（approximately 2 years）
  Adverse Events
The maximum tolerated dose and/or the recommended phase II dose of XZ120 | Course 1 （the first 3 weeks of treatment）
  Dose Finding